CLINICAL TRIAL: NCT06514131
Title: Evaluation of the Effectiveness of a Waterless Hygiene Technology for Totally Dependent Hospitalized Patients: A Randomized Controlled Study
Brief Title: Water Hygiene Versus Waterless Hygiene Technology for Totally Dependent Hospitalized Patients
Acronym: IGIENE-FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Azienda USL - IRCCS di Reggio Emilia (Unknown); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Azienda Ospedaliera, Ospedale Civile di Legnano (Other); University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Lea Godino, Principal Investigator - Research Nurse, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IGIENE-FAST
Record Dates: First submitted 2023-11-11; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Health Care Associated Infection
Keywords: hygiene
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants enrolled in the experimental arm will receive a perineal hygiene with pre-moistened wipes without water.
  Interventions: Procedure: Pre-moistened wipes
- Control group (No Intervention): Participants enrolled in the no intervention arm will receive perineal hygiene with soapy disposable knobs and water.

INTERVENTIONS:
Procedure: Pre-moistened wipes — Patients receiving the experimental treatment will have perineal hygiene performed with the pre-moistened wipes without water
  Arms: Experimental group

SUMMARY:
The aim of this randomized controlled trial is to verify whether the efficacy of perineal hygiene procedures performed in dependent patients admitted to medical or geriatric wards with pre-moistened wipes without water is higher than that found after procedures performed with disposable hand grips, soap, and water.

DETAILED DESCRIPTION:
Patients hospitalized in medicine and geriatrics wards will be admitted, both for scheduled and urgent hospitalizations. If the patient meets the study inclusion criteria, we will proceed with the description of the study, the delivery of the information form and the collection of informed consent. Only after signing the consent, the patient can be enrolled in the study. The day following enrollment, the first perineal hygiene in the morning will be performed with pre-moistened wipes without water or with disposable hand grips, soap and water depending on the study group to which the patient has been randomly assigned.

In both groups, a skin swab will be performed before and after the hygiene practice, after which the patient will leave the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age inclusive at the time of the study;
* Patients admitted to medical or geriatric wards with scheduled or urgent hospitalization;
* Hypothesis of hospitalization of at least 48 hours
* Totally dependent patients who are bedridden and unable to independently provide for their own personal hygiene.
* Patient-oriented in time and space/cognitively cooperative.
* Acquisition of written informed consent.

Exclusion Criteria:

* Patients who have performed perineal hygiene with wipes or other methods containing antiseptic solutions in the 12-24 hours preceding the execution of the swab for the bacteriological examination.
* Patients who have undergone a treatment procedure in the groin and/or perineal area that required skin antisepsis (e.g. femoral blood sampling, bladder catheter insertion, etc.).
* Patients with known allergies to one of the components of the products used.
* Patients diagnosed with dermatological pathologies.
* Patients colonized or infected with microorganisms transmissible by contact.
* Patients in bowel cleansing preparation for diagnostic procedures e therapeutic.
* Patients with diarrheal bowel.
* Patients hospitalized on Saturdays and Sundays due to the difficulty of illustrating information and acquiring informed consent since healthcare professionals are small in number.
* Patient enrolled and then transferred to another ward or discharged before 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Microbial load : effectiveness of the perineal hygiene with pre-moistened wipes | One day
  The primary objective is to verify if the effectiveness of the perineal hygiene procedures performed in hospitalized dependent patients in medicine or geriatric wards with pre-moistened wipes without water (experimental treatment) is higher than that found after the procedures performed with soapy disposable grips and water (standard treatment). Each patient will be treated with one of the two methods only once; for each patient, a total of two measurements of microbial load will be performed pre- and post-morning hygiene. Change from baseline in microbial load will be evaluated.

SECONDARY OUTCOMES:
Compare the total costs of the aids used in the two hygiene methods | One day
  Cost of materials and personnel
Compare the working times referred to the two hygiene methods | One day
  Time expressed in minutes, required for the completion of perineal hygiene for each methodology
Compare the patients' satisfaction with the two hygiene methods | One day
  Assessed by a specific ad hoc questionnaire ranging from 2 to 10 (higher scores mean a better outcome)
Compare the approval of health professionals for the two hygiene methods | One day
  Assessed by a specific ad hoc questionnaire ranging from 2 to 10 (higher scores mean a better outcome)
Examine the patient-operator concordance regarding the different aspects relating to the liking for the two hygiene methodologies | One day
  Assessed by a specific ad hoc questionnaire (list of items)

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Azienda Ospedaliera, Ospedale Civile di Legnano, Legnano, Milano
  - IRCCS AOU di Bologna, Bologna
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia
  - University of Rome Tor Vergata, Roma

IPD SHARING:
Plan to Share IPD: No